CLINICAL TRIAL: NCT06490120
Title: En Longitudinell Observationsstudie om Unga Individers Psykiska hälsa i Sverige
Brief Title: A Study on Young Individuals' Mental Health in Sweden
Acronym: UPIC
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: UU20230127
Record Dates: First submitted 2024-05-31; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Issue; Depression, Anxiety; Well-Being, Psychological
Keywords: Mental Health; Trajectories; Multimodal; Young Individuals; Ecological momentary assessment
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples, analysed for proteomics, metabolomics
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Protocol 1: Mental health is assessed over the course of 2 years, by survey on three occasions: at baseline and follow-ups at 1 and 2 years later.
  Interventions: Other: sampling method
- Protocol 2: Mental health is assessed over the course of 2 years, by survey on five occasions: at baseline and 6, 12, 18 and 24 months later.
  Interventions: Other: sampling method
- Protocol 3: Mental health is assessed over the course of 2 years, by survey on three occasions: at baseline and follow-ups at 1 and 2 years later. Additionally, a real-time data capture method, ecological momentary assessments (EMA) will be applied directly after baseline and 6, 12 and 18 months later. Participants in group 3 will asked to complete daily registrations using a selection of self-report measures during a one month period. The self-report questions will be distributed via the application with about 5 to 15 questions at a time.
  Interventions: Other: sampling method

INTERVENTIONS:
Other: sampling method — feasibility outcomes will be compared between the 3 groups

SUMMARY:
The goal of this observational study is to increase our knowledge about the mental health of young individuals and to establish a valid and comprehensive method for assessing mental health in young individuals (15-29 years) that can improve our capacity to promote mental health and address mental health problems.

The specific aims of the proposed project are: 1) To determine the extent and course of mental health in young men and women over a two-year period and discern the added value of multimodal data to assess and predict mental health problems. 2) To demonstrate the feasibility of different assessment methods of mental health in young individuals.

Participants will be able to provide:

* Survey data - mental health outcome measures are used to assess mental well-being and mental health problems, and sociodemographic and individual health data are collected to explore potential confounders with the primary outcomes.
* Behavioral testing - online/remote behavioral assessments such as approach-avoidance conflict, emotional regulation, risk-taking-attitude and cognitive tests.
* National register data - sociodemographic data including age, country of birth, education, school absence, sickness absence and income, inpatient (hospital) and outpatient specialist care, information on e.g. psychiatric conditions and pain conditions and psychiatric care and use of psychotropic medication.
* Blood-based biological marker - monitoring of about 800 biomarkers, carefully selected to target the most important metabolic pathways, including steroid-, hormone-, neurotransmitter- and lipid regulation.
* Passive data by digital phenotyping - automatically collected data from for example smartphone sensors and activity logs.
* App- and survey metadata - app usage, when a survey was opened, time taken to answer separate measures and questions, completion of full survey, and any changes made in survey responses.

Researchers will compare 3 different assessment protocols, with participants providing data at different time points, this in order to see demonstrate feasibility and methods for future studies on mental health in young individuals. Establishment of feasibility is done by collecting data on: recruitment rate, adherence and acceptance of study procedures including mode of data collection.

DETAILED DESCRIPTION:
In Sweden, reports show an increase in mental health problems of young people, in particular of young women. This increase is poorly understood, calling for more rigorous studies to clarify extent and severity of the problems, but also, to inform practices on how to adequately assess youth mental health.

The purpose of this project is to increase our knowledge about the mental health of young women and men and to establish a valid and comprehensive method for assessing mental health in young individuals that can improve our capacity to promote mental health and address mental health problems. A multimodal data approach is applied, comprising a feasibility study on methods of assessment of mental health in young individuals.

The specific aims of the proposed project are: 1) To determine the extent and course of mental health in young women and men over a two-year period and discern the added value of multimodal data to assess and predict mental health problems. 2) To demonstrate the feasibility of different assessment methods of mental health in young women and men. Establishment of feasibility is done by collecting data on: recruitment rate, adherence and acceptance of study procedures including mode of data collection.

There is a common opinion in Sweden and internationally that mental health problems have increased over the past decades. More research is needed to understand this proposed increase in mental health problems and to clarify if the reports reflect a genuine deterioration in mental health. Existing studies have been criticized for not being able to provide reliable estimates of mental health problems due to heterogeneity in study designs and limitations including lack of use of established, comprehensive measures. The national surveys that indicate a deterioration of mental health in young women in Sweden rely on reports from single questions. Although less respondent burden, the validity and reliability of using single questions to assess concepts such as anxiety and depression can be disputed. Moreover, existing studies provide cross-sectional point estimates rather than prospective time lines, which generally result in more accurate and reliable data.

Traditional methodologies with sole reliance on self-reported data to provide accurate and reliable estimates to better understand mental health of young women may not be the way forward. For instance, metabolomics biomarkers taken from for example blood or urine have gained interest for its ability to screen new and unsuspected pathways involved in psychiatric disorders, and fear conditioning and extinction protocols as well as behavioural testing of e.g. avoidance and distress tolerance have shown promise in detecting and predicting mental health. Combining self-report data with information from such other data sources presents a promising approach, yet the use of multimodal data is an understudied area in mental health research. Moreover, with the ubiquity of smartphones along with advances in technology, it is now possible to use digital devices such as smartphones to assess and track certain behaviours, which makes it possible to address some of the drawbacks of traditional assessment methods. Behavioural real-time data on e.g., participant's symptoms, functions, and social environment in nonclinical settings collected from digital devices holds considerable potential for detecting, understanding and predicting psychiatric conditions, mood disorders, and depressive symptoms.

This feasibility study consists of a prospective cohort using a multimodal data approach. The same theoretical framework, procedure, data collection and measurements apply to both Aim 1 and Aim 2.

Design Three assessment protocols will be evaluated. After baseline assessment, participants will be randomly assigned to a protocol on a 1:1:1 basis. Considering participant dropout after baseline and with an aim to include 750 young individuals per protocol, recruitment will continue until the target number of 200 young individuals per year of birth at baseline (n=3000) is reached. The proposed sample size is based on our primary feasibility outcome: complete adherence of the protocol. Assuming 90% power and alpha=0.05, at least 500 young individuals are needed to adhere to each protocol to detect a 10% statistically significant difference in adherence between protocols, e.g. 60% adherent young individuals assigned to protocol 1 and 2, who complete follow-up, compared with 50% adherent young individuals assigned to protocol 3.

Data collection Data from different modalities will be combined, including both active and passive data. Specifically, data will be collected by survey, smartphone sensor data, at-home blood sampling, behavioural tests, and register data. Most data will be administered via a study-specific app. Written (electronic) consent will be obtained before participation. For instance, a participant may consent to participation with survey data, sensor data, and behavioural tests, but not with blood sample or linkage to register data. Incentives will be offered to participants at completion of an assessment.

In protocol 1, mental health is assessed by survey on three occasions: at baseline and follow-ups at 1 and 2 years later. This design with yearly assessments is congruent with conventional methods of assessment by survey. To investigate the potential benefits as well as risks of more frequent assessments, data will be collected in the same way in protocol 2, but on five occasions: at baseline and 6, 12, 18 and 24 months later. In protocol 3, in addition to yearly assessments by survey, a real-time data capture method referred to as ecological momentary assessments (EMA) will be applied. After the baseline assessment, participants in protocol 3 will asked to complete daily registrations using a selection of self-report measures during a one-month period. The self-report questions will be distributed via the application with about 15-20 questions at a time. This EMA schedule will be repeated three times over the study period.

Data analysis plan The number of young individuals who indicate caseness (according to available scoring guides) of depressive symptoms based on survey responses will be determined to assess prevalence and developmental trajectories of self-reported mental health problems over the two-year follow-up time. Mental health profiles will be mapped with the use of information from the different types of data. The statistical techniques applied for identification of symptom patterns, relationships and determinants of mental health problems and well-being will be suited to complex longitudinal and multimodal data, such as structural equation modelling, generalized linear (mixed) models, and Bayesian modelling. To study time series of symptom occurrence clusters of longitudinally reported symptoms will be obtained by unsupervised clustering analysis.

Based on previous studies on mental health in youth, a point of reference of >20% for baseline recruitment rate will be considered feasible. Dropout analysis will target representativeness at baseline and throughout the phases of the study. At baseline, the distributions of sociodemographic data obtained by register data will be analysed between participants and nonparticipants. For identification of attrition bias, dropout analysis will consider sociodemographic register data but also analyse distributions of health outcomes from previous assessments among participants and dropouts at later stages of the study.

An adherence rate of >50% during the two-year follow-up will be considered feasible, and will be evaluated for each assessment protocol. For the EMA outcomes (protocol 3), the recording and reporting of compliance data will follow the published recommendations, including the measurement of compliance rate as number of prompts answered out of the total number of prompts delivered (compliance of ≥80% feasible) and latency (time period between when participants receive a prompt and when the EMA is answered). Based on previous survey studies on mental health in Sweden, an overall compliance of >75% will be considered feasible. A feasible acceptance rate of behaviour experiments in this heterogeneous, nonclinical population cannot be decided, but our results will clarify acceptance and completion rate for this kind of remotely delivered behavioural experiment. Based on preliminary results of the Mom2B study, an acceptance rate of >70% for access to passive data and 80% to register data will be considered feasible. Furthermore, the completion rate of each self-report measure will be calculated. Instrument guidelines will guide the analyses and interpretation, but if no guideline exists <10% internal missing per question/scale is considered feasible.

Expected outcome The prospective design allows detection of extent and severity of mental health problems in young individuals and will clarify the course of mental health during a two-year period. To clarify the added value of having more frequent assessment points to detect course of mental health is an important outcome of the present study. The results of the EMA assessments will reveal individual day-to-day variability across mental health symptoms and behaviors, expanding the knowledge of the underlying processes and dynamics of mental health. The results will demonstrate the utility of multimodal data for the assessment of mental health and show how outcomes from different data sources are interrelated. This, along with the identification of potential drawbacks of frequent assessments will guide future health assessment strategies. It also allows for data on the predictive value of health outcomes from different methods of assessment. Of particular interest is to demonstrate if multimodal data provide more comprehensive data than single data modality and to clarify if multimodal data improve precision in prediction of mental health problems.

Importantly, the results will demonstrate if an age- and sex-stratified recruitment strategy is appropriate or if selective recruitment methods are needed to obtain a representative population sample. The feasibility of collecting mental health data by self-report measures with 6-month and/or one year follow-up as well as with an EMA approach will be clarified. Results will also show if behavioural testing, passive data, blood sampling are feasible outcome tools to use as proposed.

ELIGIBILITY:
Inclusion Criteria:

* age at recruitment
* ownership of smartphone

Exclusion Criteria:

* N/A

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Men and women in the general population in Sweden aged 15-29 years at recruitment
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Generalised Anxiety Disorder (GAD-7). Swedish version. 7 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. 1 item ranging from 0 ='not at all, to 3 = 'very disturbing'. The first 7 items are summed to a sum score ranging from 0 to 21, where: 0-4 = no signs of anxiety, 5-9 = mild GAD, 10-14 = moderate GAD, 15-21 = severe GAD. Item 8 is reported as a single item where higher score means higher interference.
Change in anxiety symptoms | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Generalised Anxiety Disorder (GAD-7). Swedish version. 7 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. 1 item ranging from 0 ='not at all, to 3 = 'very disturbing'. The first 7 items are summed to a sum score ranging from 0 to 21, where: 0-4 = no signs of anxiety, 5-9 = mild GAD, 10-14 = moderate GAD, 15-21 = severe GAD. Item 8 is reported as a single item where higher score means higher interference.
Change in depressive symptoms | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Patient Health Questionnaire - 9 (PHQ-9+1), Swedish version. 9 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. The first 9 items are summed to a sum score ranging from 0 to 27, where: 0-4 = no signs of depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression. Item 10 is reported as a single item where high scores indicate high interference with daily function.
Change in depressive symptoms | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Patient Health Questionnaire - 9 (PHQ-9+1), Swedish version. 9 items ranging from 0 ='not at all', to 3 ='almost every day'. 1 item ranging from 0 ='no difficulties, to 3 = 'extreme difficulties'. The first 9 items are summed to a sum score ranging from 0 to 27, where: 0-4 = no signs of depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, 20-27 = severe depression. Item 10 is reported as a single item where high scores indicate high interference with daily function.
Change in well-being | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Well-Being Index (WHO-5). Swedish version. 5 items ranging from 0 ='at no time', to 5 ='all the time'. The 5 items are summed to a score ranging from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Change in well-being | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Well-Being Index (WHO-5). Swedish version. 5 items ranging from 0 ='at no time', to 5 ='all the time'. The 5 items are summed to a score ranging from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.

SECONDARY OUTCOMES:
Change in emotional well-being | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Mental Health Continuum Short Form (MHC-SF). Swedish version. 14 items which assesses how often a statement was true during the past two weeks, reported on a 6-point Likert scale ranging from 0 "never" to 5 "everyday". Statements include emotional, social, and psychological aspects of well-being. Items are summed, yielding a total score ranging from 0 to 70. The total scale score will be used for the assessment of overall mental well-being with higher scores indicating greater levels of positive well-being.
Change in emotional well-being | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Mental Health Continuum Short Form (MHC-SF). Swedish version. 14 items which assesses how often a statement was true during the past two weeks, reported on a 6-point Likert scale ranging from 0 "never" to 5 "everyday". Statements include emotional, social, and psychological aspects of well-being. Items are summed, yielding a total score ranging from 0 to 70. The total scale score will be used for the assessment of overall mental well-being with higher scores indicating greater levels of positive well-being.
Change in stress | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Perceived Stress Scale (PSS-10). Swedish version. 10 item ranging from 0 ='never' to 4 ='very often'. Scores for item 4, 5, 7 and 8 need to be reversed (0=4, 1=3, 2=2, 1=4) and all summed to a score ranging 0 to 40. Higher scores indicate higher level of perceived stress.
Change in stress | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Perceived Stress Scale (PSS-10). Swedish version. 10 item ranging from 0 ='never' to 4 ='very often'. Scores for item 4, 5, 7 and 8 need to be reversed (0=4, 1=3, 2=2, 1=4) and all summed to a score ranging 0 to 40. Higher scores indicate higher level of perceived stress.
Change in sleep | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: The insomnia severity index (ISI). Swedish version. The ISI comprises 7 items that assess current (i.e., preceding 2 weeks) sleep problems. The first three items evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems. Subsequent items assess current sleep problem, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and amount of worry due to the current sleep problem. Items are rated on a five-point Likert scale ('0' representing none or not at all and '4' representing very much). Total scores range from 0 to 28, with higher combined scores indicating worse insomnia severity.
Change in sleep | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: The insomnia severity index (ISI). Swedish version. The ISI comprises 7 items that assess current (i.e., preceding 2 weeks) sleep problems. The first three items evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems. Subsequent items assess current sleep problem, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and amount of worry due to the current sleep problem. Items are rated on a five-point Likert scale ('0' representing none or not at all and '4' representing very much). Total scores range from 0 to 28, with higher combined scores indicating worse insomnia severity.
Change in psychological flexibility | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: Selected items from the Multidimensional Psychological Flexibility Inventory (MPFI). Swedish version. 12 items where rate how often they experience each statement during the last 2 weeks, with responses given on a 6-point scale ranging from never true (1) to always true (6).
Change in Psychological Flexibility | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Selected items from the Multidimensional Psychological Flexibility Inventory (MPFI). Swedish version. 12 items where rate how often they experience each statement during the last 2 weeks, with responses given on a 6-point scale ranging from never true (1) to always true (6).
Change in effortful control | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: The Adult Temperament Questionnaire (ATQ). Swedish version. 19 items where Each item is rated on a 7-point Likert scale, ranging from 1 = 'extremely untrue of you' to 7 = 'extremely true of you'.
Change in effortful control | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: The Adult Temperament Questionnaire (ATQ). Swedish version. 19 items where Each item is rated on a 7-point Likert scale, ranging from 1 = 'extremely untrue of you' to 7 = 'extremely true of you'.
Change in emotion regulation | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: The Adolescents' Emotion Regulation Strategies Questionnaire-Extended (AERSQ-E). Swedish version. 23 items with each item rated on a 5-point scale, ranging from 1 = 'very rarely/never' to 5 = 'very often/always'.
Change in emotion regulation | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: The Adolescents' Emotion Regulation Strategies Questionnaire-Extended (AERSQ-E). Swedish version. 23 items with each item rated on a 5-point scale, ranging from 1 = 'very rarely/never' to 5 = 'very often/always'.
Individual health data | Baseline for Group 1, 2, 3
  Self-report: height, weight, sexual health, menstrual bleeding pattern, physical health, psychological diagnosis and treatments.
Individual health data | 6 months for Group 2
  Self-report: height, weight, sexual health, menstrual bleeding pattern, physical health, psychological diagnosis and treatments.
Individual health data | 1 year for Group 1, 2, 3
  Self-report: height, weight, sexual health, menstrual bleeding pattern, physical health, psychological diagnosis and treatments.
Individual health data | 1.5 year Group 2
  Self-report: height, weight, sexual health, menstrual bleeding pattern, physical health, psychological diagnosis and treatments.
Individual health data | 2 year for Group 1, 2, 3
  Self-report: height, weight, sexual health, menstrual bleeding pattern, physical health, psychological diagnosis and treatments.
Health behaviours | Baseline for Group 1, 2, 3
  Self-report: physical activity, habits related to smoking, alcohol use, caffein, food and fluid intake. Social media use and leisure time.
Health behaviours | 6 months for Group 2
  Self-report: physical activity, habits related to smoking, alcohol use, caffein, food and fluid intake. Social media use and leisure time.
Health behaviours | 1 year for Group 1, 2, 3
  Self-report: physical activity, habits related to smoking, alcohol use, caffein, food and fluid intake. Social media use and leisure time.
Health behaviours | 1.5 year Group 2
  Self-report: physical activity, habits related to smoking, alcohol use, caffein, food and fluid intake. Social media use and leisure time.
Health behaviours | 2 year for Group 1, 2, 3
  Self-report: physical activity, habits related to smoking, alcohol use, caffein, food and fluid intake. Social media use and leisure time.
Sociodemographic data | Baseline for Group 1, 2, 3
  Self-report: country of birth, gender, sexual identity, living situation, employment, education.
Sociodemographic data | 6 months for Group 2
  Self-report: country of birth, gender, sexual identity, living situation, employment, education.
Sociodemographic data | 1 year for Group 1, 2, 3
  Self-report: country of birth, gender, sexual identity, living situation, employment, education.
Sociodemographic data | 1.5 year Group 2
  Self-report: country of birth, gender, sexual identity, living situation, employment, education.
Sociodemographic data | 2 year for Group 1, 2, 3
  Self report: country of birth, gender, sexual identity, living situation, employment, education.
Social factors | Baseline for Group 1, 2, 3
  Self-report: sense of community and belonging, and experience of violence and harassment
Social factors | 6 months for Group 2
  Self-report: sense of community and belonging, and experience of violence and harassment
Social factors | 1 year for Group 1, 2, 3
  Selfreport: sense of community and belonging, and experience of violence and harassment
Social factors | 1.5 year Group 2
  Self-report: sense of community and belonging, and experience of violence and harassment
Social factors | 2 year for Group 1, 2, 3
  Self-report: sense of community and belonging, and experience of violence and harassment
Explorative identification of biomarkers | Baseline for Group 2, 3
  Optional at home blood sample, extraction and analysis of about 800 biomarkers and ratios of metabolic pathways, including steroid-, hormone-, neurotransmitter- and lipid regulation
Explorative identification of biomarkers | 6 months for Group 2, 3
  At home blood sample, extraction and analysis of about 800 biomarkers and ratios of metabolic pathways, including steroid-, hormone-, neurotransmitter- and lipid regulation
Behavioral test, approach-avoidance conflict | Baseline for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as approach-avoidance conflict.
Behavioral test, emotional regulation | Baseline for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as emotional regulation.
Behavioral test, risk-taking | Baseline for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as risk-taking.
Behavioral test, influence of ambiguity | Baseline for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as influence of ambiguity.
Behavioral test, approach-avoidance conflict | 1 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as approach-avoidance conflict.
Behavioral test, emotional regulation | 1 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as emotional regulation.
Behavioral test, risk-taking | 1 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as risk-taking.
Behavioral test, influence of ambiguity | 1 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as influence of ambiguity.
Behavioral test, approach-avoidance conflict | 2 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as approach-avoidance conflict.
Behavioral test, emotional regulation | 2 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as emotional regulation.
Behavioral test, risk-taking | 2 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as risk-taking.
Behavioral test, influence of ambiguity | 2 year for Group 1, 2, 3
  Data from online, remote behavioural tests. Measures of basic psychological mechanisms of importance for mental health such as influence of ambiguity.
Change in curiosity | Baseline, 1 year, 2 year for Group 1 and 3
  Self Report: Five-Dimensional Curiosity Scale Revised (5DCR). Swedish version. 7 selected items from Five-Dimensional Curiosity Scale Revised (5DCR). 7-point scale ranging from 1 = 'does not describe me' to 7 = 'describes me completely'.
Change in curiosity | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: Five-Dimensional Curiosity Scale Revised (5DCR). Swedish version. 7 selected items from Five-Dimensional Curiosity Scale Revised (5DCR). 7-point scale ranging from 1 = 'does not describe me' to 7 = 'describes me completely'.
Change in perceived meaningfulness of leisure | Baseline, 1 year, 2 year for Group 1 and 3
  Self-report: 1 item. 4-point scale ranging from not at all meaningful (0) to absolutely meaningful (4).
Change in perceived meaningfulness of leisure | Baseline, 6 months, 1 year, 1.5 years, 2 year for Group 2
  Self-report: 1 item. 4-point scale ranging from not at all meaningful (0) to absolutely meaningful (4).

OTHER OUTCOMES:
Feasibility, Recruitment | Baseline
  Number of individuals needed to be approached to include desired number of participants at baseline in every age group.
Feasibility, Number of participants that adhere to each assessment protocol (group) | Throughout the 2 year study period
  Number of participants that adhere to each assessment protocol (group). For participants' in group 3, number of participants that adhere to the EMA will be registered for each monitoring period.
Feasibility, Acceptance of study | Throughout the 2 year study period
  Number of individuals that consent to participate in the study.
Feasibility, Acceptance of optional parts of study | Throughout the 2 year study period
  Number of individuals that consent to participate in any of the optional data collection procedures of the study.
Feasibility, Completion rates | Throughout the 2 year study period
  Completion rates for the data collection procedures will be assessed. Completion rate means the ratio of the number of participants who complete a data procedure to the total number of participants eligible.
Feasibility, Missing data | Throughout the 2 year study period
  Amount of missing values in survey responses.
National registry data, Health care episodes in inpatient (hospital) | Pre-baseline and continuous over the 2 year study period
  Data on health care episodes in inpatient (hospital).
National registry data, Outpatient specialist care | Pre-baseline and continuous over the 2 year study period
  Data on outpatient specialist care, including psychiatric care.
National registry data, Psychiatric conditions | Pre-baseline and continuous over the 2 year study period
  Data on psychiatric conditions.
National registry data, Pain conditions | Pre-baseline and continuous over the 2 year study period
  Data on pain conditions.
National registry data, Co-morbidity of psychiatric and pain conditions | Pre-baseline and continuous over the 2 year study period
  Data on co-morbidity of psychiatric and pain conditions.
National registry data, Psychotropic medication | Pre-baseline and continuous over the 2 year study period
  Use of psychotropic medication.
National registry data, School absence | Pre-baseline and continuous over the 2 year study period
  Data on school absence.
Smartphone sensor data, Internet usage | Continuous over the 2 year study period
  Sensor data on internet usage.
Smartphone sensor data, Reachability | Continuous over the 2 year study period
  Sensor data on reachability (if connected or not to cellular network, Wi-Fi).
Smartphone sensor data, General smartphone activity | Continuous over the 2 year study period
  Sensor data on general smartphone activity (processor use (%))
Smartphone sensor data, Internet activity | Continuous over the 2 year study period
  Sensor data include on internet activity (kb/s).
Smartphone sensor data, Internet availability | Continuous over the 2 year study period
  Sensor data on internet availability.
Smartphone sensor data, Charger use | Continuous over the 2 year study period
  Sensor data on charger use.
Smartphone sensor data, Geographical movement patterns | Continuous over the 2 year study period
  Sensor data geographical movement patterns (measured with location services (GPS) and the accelerometer.
Survey and app metadata, Survey opened | Continuous over the 2 year study period
  App usage: when a survey was opened.
Survey and app metadata, Time to answer separate measures and questions | Continuous over the 2 year study period
  App usage: time taken to answer separate measures and questions.
Survey and app metadata, Completion of full survey | Continuous over the 2 year study period
  App usage: completion of full survey.
Survey and app metadata, Changes made in survey responses | Continuous over the 2 year study period
  App usage: any changes made in survey responses.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden